CLINICAL TRIAL: NCT06032065
Title: Sequential Multiple Assessment Randomized Trial of Exercise for PAD: SMART Exercise for Peripheral Artery Disease: The SMART PAD Trial
Brief Title: SMART Exercise for PAD
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Mary McDermott, Jeremiah Stamler Professor of Medicine, Northwestern University
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STU00218112
Record Dates: First submitted 2023-05-22; First posted 2023-09-11 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Peripheral Arterial Disease; Aging; Peripheral Vascular Diseases; Walking, Difficulty
Keywords: behavior change; patient reported outcome measure
MeSH Terms: conditions — Peripheral Arterial Disease; Peripheral Vascular Diseases; Mobility Limitation

STUDY DESIGN:
Intervention Model Description: The investigators will use a 2 x 2 factorial design to address two major barriers to achieving benefits from exercise therapy for PAD: First, guideline recommendations for supervised exercise therapy (SET) as first line therapy for PAD. Second, the inability of exercise therapy to eliminate PAD-related disability in most people with PAD. In this 2 x 2 factorial design, participants will be randomized to one of four groups for 12 weeks: Supervised treadmill exercise + nitrate rich beetroot juice; supervised treadmill exercise + placebo, home-based walking exercise + nitrate rich beetroot juice, home-based walking exercise + placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: For the beetroot juice vs. placebo comparison, this will be a double blinded study where both the participant and the people collecting data will be blinded. For the supervised exercise vs. home-based exercise comparison, the participant and investigator will not be blinded, but the outcomes assessor will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Supervised treadmill exercise + nitrate rich beetroot juice (Experimental): This group will be participating in Supervised Treadmill Exercise and drinking nitrate rich beetroot juice for 12 weeks.
  Interventions: Behavioral: Supervised Treadmill Exercise; Dietary Supplement: Nitrate-rich beetroot Juice
- Supervised treadmill exercise + placebo (Placebo Comparator): This group will be participating in Supervised Treadmill Exercise and drinking placebo beetroot juice with nitrate removed for 12 weeks.
  Interventions: Behavioral: Supervised Treadmill Exercise
- Home-based walking exercise + nitrate rich beetroot juice (Experimental): This group will be participating in Home-Based Exercise and drinking nitrate rich beetroot juice for 12 weeks.
  Interventions: Behavioral: Home-Based Exercise; Dietary Supplement: Nitrate-rich beetroot Juice
- Home-based walking exercise + placebo (Placebo Comparator): This group will be participating in Home-Based Exercise and drinking placebo beetroot juice with nitrated removed for 12 weeks.
  Interventions: Behavioral: Home-Based Exercise

INTERVENTIONS:
Behavioral: Supervised Treadmill Exercise — This is a 12 week intervention where participants will walk for exercise 3 times a week on a treadmill at a center while being supervised by healthcare personnel.
  Arms: Supervised treadmill exercise + nitrate rich beetroot juice; Supervised treadmill exercise + placebo
Behavioral: Home-Based Exercise — This is a 12 week intervention where participants will walk at home for exercise with guidance from a study coach. They will have 4 in person visits in the first four weeks and then have weekly phone calls in the last 8 weeks of the intervention with their coach.
  Arms: Home-based walking exercise + nitrate rich beetroot juice; Home-based walking exercise + placebo
Dietary Supplement: Nitrate-rich beetroot Juice — Participants will drink one shot of nitrate rich beet-root juice twice daily for 12 weeks.
  Arms: Home-based walking exercise + nitrate rich beetroot juice; Supervised treadmill exercise + nitrate rich beetroot juice

SUMMARY:
Supervised exercise therapy (SET), consisting of treadmill exercise conducted three times weekly at a center while supervised by healthcare personnel, is first line therapy for people disabled by lower extremity peripheral artery disease (PAD). However, travelling three times/week to a center for SET is burdensome. Compared to SET, home-based exercise is more accessible and less burdensome. Yet, evidence-based guidelines recommend SET over home-based exercise for PAD. Walking exercise is first line therapy to improve walking distance for PAD, but it does not eliminate ischemic leg symptoms in most people with PAD. The investigators' work and that of others showed that nitrate-rich beetroot juice, which increases plasma nitrite, limb perfusion, and skeletal muscle function, significantly improved exercise tolerance and reduced non-response to exercise in people with and without PAD. The investigators will use a 2 x 2 factorial design to address two major barriers to achieving benefits from exercise therapy for PAD: First, guideline recommendations for supervised exercise therapy (SET) as first line therapy for PAD. Second, the inability of exercise therapy to eliminate PAD-related disability in most people with PAD. Participants will be randomized to one of four groups for 12 weeks: Supervised treadmill exercise + nitrate rich beetroot juice; supervised treadmill exercise + placebo, home-based walking exercise + nitrate rich beetroot juice, home-based walking exercise + placebo.

DETAILED DESCRIPTION:
Supervised exercise therapy (SET), consisting of treadmill exercise conducted three times weekly at a center while supervised by healthcare personnel, is first line therapy for people disabled by lower extremity peripheral artery disease (PAD). However, travelling three times/week to a center for SET is burdensome. As of 2018, only 1.3% of patients with Medicare and symptomatic PAD had enrolled in SET. Compared to SET, home-based exercise is more accessible and less burdensome. Yet, evidence-based guidelines recommend SET over home-based exercise for PAD. In 2021, the investigators reported that a home-based exercise intervention that incorporated behavioral methods significantly improved six-minute walk in PAD, compared to an attention control group. But no randomized trials have compared SET to a home-based exercise intervention that incorporated behavioral change methods in PAD. However, 45% of people with PAD do not meaningfully respond to exercise interventions, defined as failure to improve six-minute walk by > 20 meters. This phenomenon occurs for both supervised and home-based exercise. The investigators' work and that of others showed that nitrate-rich beetroot juice, which increases plasma nitrite, limb perfusion, and skeletal muscle function, significantly improved exercise tolerance and reduced non-response to exercise in people with and without PAD. Therefore, the investigators will use a 2 x 2 factorial design to address two major barriers to achieving benefits from exercise therapy for PAD: First, guideline recommendations for supervised exercise therapy (SET) as first line therapy for PAD. Second, the inability of exercise therapy to eliminate PAD-related disability in most people with PAD. In this 2 x 2 factorial design, participants will be randomized to one of four groups for 12 weeks: Supervised treadmill exercise + nitrate rich beetroot juice; supervised treadmill exercise + placebo, home-based walking exercise + nitrate rich beetroot juice, home-based walking exercise + placebo.

ELIGIBILITY:
Inclusion Criteria:

First, all participants will be age 50 and older. Second, all participants will have PAD. PAD will be defined as either:

1. An ABI <= 0.90 at baseline.
2. Vascular lab evidence of PAD (such as a toe brachial pressure less than or equal to 0.70 or an ankle brachial index less than or equal to 0.90), or angiographic evidence of PAD defined as at least 70% stenosis of an artery supplying the lower extremities.
3. An ABI of >0.90 and <1.00 who experience a 20% or greater drop in ABI in either leg after the heel-rise test.

Exclusion Criteria:

1. Above- or below-knee amputation
2. Limb-threatening ischemia defined as an ABI <0.40 with symptoms of rest pain
3. Wheelchair confinement or requiring a walker to ambulate
4. Walking is limited by a condition other than PAD
5. Current foot ulcer on bottom of foot
6. Unwilling to drink beetroot juice
7. Unwilling to accept randomization into either group (home based exercise or supervised exercise)
8. Planning to engage in new walking exercise outside of the study or unwilling to refrain from new walking exercise activity during the trial.
9. Already exercising at a level consistent with exercise intervention.
10. End-stage kidney disease (ESKD) associated with the need for dialysis.
11. Planned major surgery, coronary or leg revascularization during the next six months
12. Major surgery, coronary or leg revascularization or major cardiovascular event in the previous three months
13. Major medical illness including lung disease requiring oxygen, Parkinson's disease, a life-threatening illness with life expectancy less than six months, or cancer requiring treatment in the previous two years. [NOTE: potential participants may still qualify if they have had treatment for an early stage cancer in the past two years and the prognosis is excellent. Participants who require oxygen only at night may still qualify.]
14. Mini-Mental Status Examination (MMSE) score < 23 or dementia. However, if the MMSE is < 23 and the Principal Investigator evaluation determines that the lower score is related to language barriers or education level, the Principal Investigator has discretion to allow a participant with MMSE < 23 to participate, as appropriate.
15. Allergy to beetroot juice
16. Currently consuming beetroot juice or oral nitrate or nitrite, or a beetroot supplement, and/or unwilling to avoid these during study participation. Participants currently consuming one cup of beets daily will be asked to discontinue beet ingestion for 30 days before baseline testing and throughout the clinical trial. If the potential participant is unwilling to refrain from daily beet consumption of one cup or more, they will not be eligible for the clinical trial.
17. Unstable angina
18. Abnormal baseline stress test without subsequent clearance for exercise by physician
19. Non-English speaking. The SMART PAD interventions are delivered by interventionists who do not speak non-English languages. The integrity of the clinical trial requires clear and effective communication for data collection and intervention delivery. The trial does not have staff members who are fluent in non-English languages, nor does it have the ability to translate all study materials into other languages.
20. Participation in or completion of a clinical trial in the previous three months. [NOTE: after completing a stem cell or gene therapy intervention, participants will become eligible after the final study follow-up visit of the stem cell or gene therapy study so long as at least six months have passed since the final intervention administration. After completing a supplement or drug therapy (other than stem cell or gene therapy), participants will be eligible after the final study follow-up visit as long as at least three months have passed since the final intervention of the trial.] Participants in a study that involved up to three single doses of nitrate-rich beetroot juice administered on separate days may participate if a month has passed since their last dose of nitrate-rich beetroot juice.
21. Visual impairment that limits walking ability.
22. Baseline blood pressure <100/45.
23. Participation in a supervised treadmill exercise program or cardiac rehabilitation program in previous three months.
24. Using a mouthwash containing chlorhexidine or cetylpyridinium chloride or a mouthwash determined to be bactericidal and unwilling to discontinue.
25. In addition to the above criteria, investigator discretion will be used to determine if the trial is unsafe or not a good fit for the potential participant.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2023-09-08 (Actual); Primary Completion 2028-11-01 (Estimated); Study Completion 2029-03-31 (Estimated)

PRIMARY OUTCOMES:
Six-Minute Walk Distance | Measured at baseline and 12 week follow-up
  Change in six-minute walk distance

SECONDARY OUTCOMES:
Walking Impairment Questionnaire (WIQ) Distance Score | measured at baseline and 12 weeks
  WIQ distance score - Range 0-100, 100 is best.
PROMIS Mobility Questionnaire Score | measured at baseline and 12 weeks
  PROMIS mobility score from administered PROMIS questionnaire. Score range is from zero to infinity and a higher score means a better outcome.
20-meter Improvement in Six-Minute Walk Distance | measured at 12 weeks
  Meaningful response to exercise interventions
Step Count | measured at baseline and 12 weeks
  Step count measured over seven days with the FITBIT
Six-Minute Walk Distance | Measured at baseline and 24-week follow up
  Change in six-minute walk distance

OTHER OUTCOMES:
Physical Activity Step Count | Measured at baseline and 24 weeks
  Step count measured over seven days with FITBIT
Physical activity distance | Measured at baseline and 24 weeks.
  Physical activity distance measured over seven days with FITBIT
Short physical performance battery (SPPB) | measured at baseline and 12 weeks
  SPPB range, range 0-12, 12-best
Walking Impairment Questionnaire (WIQ) Stair Climbing Score | measured at baseline and 12 weeks
  WIQ stair climbing score from administered WIQ, range 0-100, 100 is best.
Walking Impairment Questionnaire (WIQ) Walking Speed Score | measured at baseline and 12 weeks
  WIQ walking speed score from administered WIQ, range 0-100, 100 is best
Walking Impairment Questionnaire (WIQ) Stair Climbing Score | measured at baseline and 24 weeks
  WIQ stair climbing score from administered WIQ, range 0-100, 100 is best
Walking Impairment Questionnaire (WIQ) Walking Speed Score | measured at baseline and 24 weeks
  WIQ walking speed score from administered WIQ, range 0-100, 100 is best
Short physical performance battery (SPPB) | measured at baseline and 24 weeks
  SPPB range, range 0-12, 12-best
Physical Activity Total Distance | Measured at baseline and 12 weeks
  Distance walked over seven days measured with FITBIT

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - University of Minnesota, Minneapolis, Minnesota